CLINICAL TRIAL: NCT00797576
Title: Detection of Left Atrial Appendage Thrombus in Patients Referred For Cardioversion: Comparative Analysis of Cardiac Magnetic Resonance Imaging and Transesophageal Echocardiogram
Brief Title: Detection of Left Atrial Appendage (LAA) Thrombus: Comparison of Cardiac Magnetic Resonance Imaging and Transesophageal Echocardiogram
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Gundersen Lutheran Health System (Other)
Responsible Party: Raju G Ailiani, MD, Gundersen Lutheran Helath system
Other Study IDs: 2-07-05-001
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-08

CONDITIONS: Left Atrial Appendage Thrombi
Keywords: left atrial appendage thrombi; transesophageal echocardiogram; cardiac magnetic resonance imaging; atrial fibrillation; cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1/Cases: Subjects whom had cardioversion aborted due to LAA thrombus or suspicion of LAA thrombus on TEE.
- 2/Controls: Subjects with underlying atrial fibrillation undergoing elective TEE as clinically indicated for any reason.

SUMMARY:
The purpose of this study is to compare Cardiac Magnetic Resonance (CMR) Imaging with transesophageal echocardiography (TEE) in detecting the presence of LAA thrombi in men and women with atrial fibrillation presenting for cardioversion.

DETAILED DESCRIPTION:
The identification of left atrial appendage (LAA) thrombus prior to cardioversion for patients with atrial fibrillation is crucial. LAA thrombus can be a frequent cause of cerebral stroke or peripheral embolism post cardioversion, and anticoagulation therapy is required in these instances to prevent cerebral events and avoid embolization. To date, TEE has been considered the clinical reference in detection of LAA thrombi with high diagnostic accuracy. However, diagnosis and size estimation of LAA thrombi remains challenging due to the complex anatomy of the LAA, and transesophageal echocardiography (TEE) is considered a semi-invasive procedure. To date, there have been few comparative studies involving TEE and cardiac magnetic resonance (CMR) imaging, and the results have been conflicting. With newer CMR Imaging techniques now available, we hypothesize that comparable results will be achieved in detecting LAA thrombus in subjects using a less invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation

Exclusion Criteria:

* ICDs
* pacemakers
* intracranial clips
* intracranial stimulator devices
* insulin pumps
* intra ocular metal foreign bodies
* cochlear implants
* LAA amputation as part of CABG and/or valve surgery
* GFR < 60 mL/min

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study cases will consist of subjects referred for TEE prior to cardioversion who are found to have LAA thrombus present. Control subjects will be patients referred for TEE with chronic atrial fibrillation that will not be undergoing cardioversion. All subjects will be patients from our facility, Gundersen Lutheran Health System, La Crosse, WI.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy values for CMR Imaging for detection of LAA thrombus. (sensitivity, specificity, negative predictive value, and positive predictive value) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Raju G Ailiani, MD, Principal Investigator — Gundersen Lutheran Health System; Vicki L McHugh, MS, Study Director — Gundersen Lutheran Medical Foundation
Locations (1):
- Gundersen Lutheran Health System, La Crosse, Wisconsin, United States

REFERENCES:
- [Background] Bjerkelund CJ, Orning OM. The efficacy of anticoagulant therapy in preventing embolism related to D.C. electrical conversion of atrial fibrillation. Am J Cardiol. 1969 Feb;23(2):208-16. doi: 10.1016/0002-9149(69)90068-x. No abstract available. PMID 4180019
- [Background] Henry WL, Morganroth J, Pearlman AS, Clark CE, Redwood DR, Itscoitz SB, Epstein SE. Relation between echocardiographically determined left atrial size and atrial fibrillation. Circulation. 1976 Feb;53(2):273-9. doi: 10.1161/01.cir.53.2.273. PMID 128423
- [Background] Stein B, Halperin JL, Fuster V. Should patients with atrial fibrillation be anticoagulated prior to and chronically following cardioversion? Cardiovasc Clin. 1990;21(1):231-47; discussion 248-9. No abstract available. PMID 2199050
- [Background] Paydarfar D, Krieger D, Dib N, Blair RH, Pastore JO, Stetz JJ Jr, Symes JF. In vivo magnetic resonance imaging and surgical histopathology of intracardiac masses: distinct features of subacute thrombi. Cardiology. 2001;95(1):40-7. doi: 10.1159/000047342. PMID 11385191
- [Background] Barkhausen J, Hunold P, Eggebrecht H, Schuler WO, Sabin GV, Erbel R, Debatin JF. Detection and characterization of intracardiac thrombi on MR imaging. AJR Am J Roentgenol. 2002 Dec;179(6):1539-44. doi: 10.2214/ajr.179.6.1791539. PMID 12438051
- [Background] Ohyama H, Mizushige K, Hosomi N. Magnetic resonance imaging of left atrial thrombus. Heart. 2002 Sep;88(3):233. doi: 10.1136/heart.88.3.233. No abstract available. PMID 12181211
- [Background] Ohyama H, Hosomi N, Takahashi T, Mizushige K, Osaka K, Kohno M, Koziol JA. Comparison of magnetic resonance imaging and transesophageal echocardiography in detection of thrombus in the left atrial appendage. Stroke. 2003 Oct;34(10):2436-9. doi: 10.1161/01.STR.0000090350.73614.0F. Epub 2003 Sep 11. PMID 12970519
- [Background] Mohrs OK, Nowak B, Petersen SE, Welsner M, Rubel C, Magedanz A, Kauczor HU, Voigtlaender T. Thrombus detection in the left atrial appendage using contrast-enhanced MRI: a pilot study. AJR Am J Roentgenol. 2006 Jan;186(1):198-205. doi: 10.2214/AJR.04.1504. PMID 16357402
- [Background] Saksena S, Sra JS, Jordaens L, et al. Intracardiac Echocardiography-Guided Cardioversion Helps Interventional Procedures (ICE-CHIP) trial. Heart Rhythm Society 2007 Scientific Sessions; May 11, 2007; Denver, CO. Late Breaking clinical Trials II.